CLINICAL TRIAL: NCT02899403
Title: Neurophysiological Correlates of Cognitive Tasks in Healthy Volunteers -A Pilot Study WP3 P003
Brief Title: Neurophysiological Correlates of Cognitive Tasks in Healthy Volunteers -WP3 P003
Acronym: PharmacogWP3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013_45; 2015-A00046-43 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-09-01; First posted 2016-09-14 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Alzheimer Disease; ELECTROENCEPHALOGRAPHIC VARIANT PATTERN 1 (Disorder)
Keywords: Cognitive Tasks; Mild Cognitive Impairment; Neurophysiological Correlates; Healthy Volunteers
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy subjects (Experimental)
  Interventions: Other: Rapid Visual Information Processing (RVIP) test

INTERVENTIONS:
Other: Rapid Visual Information Processing (RVIP) test — Rapid Visual Information Processing is a measure of sustained attention.

SUMMARY:
In the perspective to better evaluate the efficacy of new treatment strategies for Alzheimer disease (AD), it appears important to develop experimental paradigms to precisely measure cognitive endpoints/biomarkers that may be used in healthy volunteers as tools to validate drug efficacy profile.

The use of Electroencephalography (EEG) may be, therefore, a good candidate. The purpose of the present study is to use EEG to more precisely explore cognitive processes in healthy subjects, with a particular interest in episodic and working memory functions that are usually altered in both AD and Mild Cognitive Impairment (MCI) as well as to better understand underlying neural mechanisms involved in these processes.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* In good health on the basis of the medical interview (medical history, symptoms), the physical examination and vital signs
* Non smoker and with no history of drug or alcohol abuse
* Without chronic treatment
* With normal hearing and normal vision including color (with correction)
* French speaker and able to understand the test instructions
* Has provided written informed consent
* Able to read and understand the Information Form and comply with the protocol instructions and restrictions

Exclusion Criteria:

* Cognitive impairment (MoCA < 26)
* Cognitive complaint (MacNair Scale > 15)
* History of brain disease (severe brain trauma, stroke, cerebral tumor…) or current cerebral disease
* Major medical or surgical history
* Current chronic disease
* Vascular or metabolic risk factor
* History or current mental disease or addiction (MINI)
* Family history of young onset dementia
* Family history of chronic or severe neurological or mental disease (first degree relatives)
* In the opinion of the investigator, is unlikely to comply with the study protocol or is unsuitable for any other reason
* Participates to another clinical trial or is still being within a washout period of a previous clinical trial
* Already exposed to cognitive tests used in this study.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-19 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
EEG spectral power during RVIP task as compared to resting state | within 7 days after inclusion ( session1)
  The Rapid Visual Information Processing (RVIP®) is a test of sustained attention and has proved useful in many studies in which drugs are used to help develop a disease model. It is sensitive to dysfunction in the parietal and frontal lobe areas of the brain

SECONDARY OUTCOMES:
EEG spectral power during PRM task as compared to resting state | within 7 days after inclusion ( session1)
  the Pattern Recognition Memory (PRM®) is a test assessing visual recognition memory, considered as a sensitive measure of medial temporal areas dysfunction. It is a useful tool for assessing patients with MCI and AD
RVIP latency of responses | within 7 days after inclusion ( session1) and within 7days after session 1 (=session2)
PRM number of errors | within 7 days after inclusion ( session1) and within 7 days after session 1 (=session2)
PRM latency of responses | within 7 days after inclusion (=session1) and within 7 days after session 1 (=session2)
difference between session 2 and session 1 EEG Spectral power during RVIP task | at 7 days after session 1

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Deplanque, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Cardiologique, CIC, Lille, France

IPD SHARING:
Plan to Share IPD: No